CLINICAL TRIAL: NCT03647826
Title: Mind Power - A CBT Based Program for Adolescents Aimed at Developing Coping Skills
Brief Title: Mind Power - A CBT Based Program for Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2510
Record Dates: First submitted 2018-07-17; First posted 2018-08-27 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Mental Depression; Mental Stress; Mental Health Wellness 1
Keywords: youth mental health; mental health prevention; empowerment
MeSH Terms: conditions — Depression; Stress, Psychological; Empowerment

STUDY DESIGN:
Intervention Model Description: Mind Power Intervention Group 1 starts in the beginning of the school semester, and Mind Power Intervention Group 2 functions as a Control Group until it starts six months after Group 1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mind Power Intervention Group 1 (Experimental): Entire school classes will be randomly divided into two interventions (Mind Power Intervention Group 1 or Mind Power Intervention Group 2). The content in the two interventions are exactly the same, except the time when they are conducted.
  The first arm is the Mind Power Intervention Group 1. This intervention is the first and starts in September 2018 and last for 10 weeks.
  Interventions: Behavioral: Mind Power Intervention
- Mind Power Intervention Group 2 (Experimental): The second arm is the Mind Power Intervention Group 2. This arm starts the intervention in January 2019 (six months later than Group 1). Group 2 function as a Control Group.
  The Experiment containes arm 1 and arm 2; With an delayed intervention design.
  Interventions: Behavioral: Mind Power Intervention

INTERVENTIONS:
Behavioral: Mind Power Intervention — The intervention has a total sample of 110 schoool classes, which are devided in two arms: Mind Power Intervention Group 1 or Mind Power Intervention Group 2

SUMMARY:
The purpose of this study is to strengthen school achievement and positive mental health, and to prevent and reduce school dropout and mental distress among high school students. The researchers will scale up techniques that have already been proven highly effective in preventing common mental disorders (depression, anxiety) in high risk groups (indicated and selective prevention). The researchers will disseminate these techniques to entire first year classes of high school students irrespective of risk factors (universal prevention). The study will report whether universal delivery in school of "Mind Power" - a Cognitive Behaviour Therapy (CBT) based programme - will strengthen school grades, self-efficacy, self-esteem, self-regulation, mental perceptions and well-being, and prevent and reduce school dropout, and symptoms of anxiety and depression. In addition the researchers will analyse whether such universal delivery prevents more mental distress, and is more cost-effective than when it is delivered only to those at high risk for school failure, dropout, or mental distress.

DETAILED DESCRIPTION:
Mind power (MTE) is a modification of the Coping With Depression (CWD) course (Lewinsohn, Weinstein, & Alper, 1970; Lewinsohn, Antonuccio, Steinmetz, & Teri, 1984). CWD is by far the most studied psycho-educational intervention (Cuijpers, Muños, Clark., & Lewinsohn, 2009). No other study has, however, tested these aims on a version of CWD. MTE is "The Adolescent Coping with Depression Course (ACDC)" (Børve, 2012). In Norwegian: "Depresjonsmesting for ungdom (DU)" and the newest version is "Mestringskurs for ungdom -DU". (The name "ACDC" has been changed to "MTE" in this project to capture the target group).

In Norway, unlike physical health training (e.g. gymnastics), mental skills training (e.g. psychological techniques in CBT) is normally reserved for individuals in treatment or at risk for developing mental disorders. However, especially in Australia and USA, universal mental skills training programmes in schools have shown positive long-term effects (e.g. Harden et al., 2001; Wells, Barlow., & Stewart-Brown, 2003).

The researchers will address how innovative research may contribute to the development of high quality education in Norway, and how to strengthen adolescents' resilience and empowerment in order to meet the challenges in society and work life. If the results in our project are positive, this project may have great impact on policy making in the areas of both education and public mental health.

Background. Why promote mental health and prevent ill-health? Depression costs society more than any other illness (Helsedirektoratet, 2015) and is one of the greatest contributors to burden of disease in Norway (Folkehelseinstituttet, 2016). Twelve per cent of both boys and girls in Norway report that they experience symptoms of depression (NOVA, 2014). Up to 80% of adolescents with mental health problems do not receive any treatment (Essau; 2005; Zachrisson, Rödje & Mykletun, 2006). Individuals (especially boys) in need of help can be reluctant to contact the mental health system because of stigma associated with mental health problems (Gulliver, Griffiths & Christensen, 2010). Universally providing mental health skills in schools to enhancing young people's social and emotional skills may compensate for this.

Dropouts from high School. Approximately 30% of adolescents in Norway do not complete high school. Approximately one third who drop out end up on disability benefit due to mental illness, mainly depression (Øverland, Glozier, Krokstad, & Mykletun, 2007; Sikveland, 2013). Internalizing problems (anxiety and depression) seems to affect dropout significantly (Melkevik et al., 2016). This has severe consequences for later work abilities, socioeconomic status and economic support (disability pensions) (Falch & Nyhus, 2011; Bergslie 2013). Because of the relationship between school motivation, mental health and academic achievements, it may be important to include all adolescents (Masten et al., 2005; Gustavsson et al., 2010).

Reduce social differences. Adolescents with multicultural backgrounds seek less help from the mental health system (Guribye & Sam, 2008). Individuals without higher education receive less help from specialists (Jensen, 2009; Mykletun, Skogen, & Knudsen, 2010). These groups may benefit from mental health skills taught in high schools, independently of socio-economic background. If the MTE intervention works, fewer adolescents may dropout from school.

Initiatives in Schools. Reviews of program evaluations show that interventions designed to promote young people's cognitive, behavioral, emotional and social development can successfully enhance skills associated with mental wellbeing (Browne, 2004; Keleher & Armstrong, 2005; Ball, 2010). There are several examples on mental skills training, such as the Friends programme, which has shown positive findings (Barrett, Farrell, Ollendick., & Dadds, 2006), along with the online CBT-programme MoodGym (Calear, Christensen, Mackinnon, Griffiths., & O'Kearney, 2009). However, most of the mental skills programs address adolescents with symptoms of anxiety and depression, or at risk of developing mental illnesses (e.g. Arnarson & Craighead, 2009).

Several mental health progammes have been evaluated in Norwegian schools; e.g. "Alle har en psykisk helse", "Zippys venner", "Ungdom møter ungdom (STEP)", "Venn1.no" (Aune & Stiles, 2009; Andersson et al., 2009; Arnesen, Breivik, Johnsen; 2005; Mishara, Ystgaad, 2006). However, these programmes are aimed mainly at teaching children about general mental health, not at teaching mental health skills universally in the classroom.

Why universal dissemination? Adolescent Coping with Depression Course (ACDC) has previously been tested on adolescents at risk for depression in a clinical setting, with positive effects (Garvik, Idsoe & Bru, 2013). However, as the prevention guru Geoffrey Rose stated: "If disease risk is widespread, measures that decrease risk for everyone are more effective in reducing the burden of disease than a 'high-risk' approach, in which measures are targeted only to those individuals with a substantially increased risk for disease." Because: "If disease rates rise continuously with higher levels of exposure to the risk factor, the larger number of people with a small elevation in risk will usually contribute more disease cases to the total burden of disease than the smaller number of people exposed to a high risk" (Rose, 2008). Rose's prevention paradigm has been proven valid on physical health by Mackenbach et al. (2012) and promising on mental health by Brugha et al. (2011). Neither CWD or ACDC have ever been tested on a non-clinical classroom sample aimed at health promotion. Because depression among young people is widespread, the researchers expect Rose's paradigm also to be valid on adolescent common mental disorder and disseminate MTE universally.

Cognitive behaviour theory (CBT). "Mental Techniques in Every-day life (MTE)" is an adaption of the "Adolescent Coping with Depression Course (ACDC) " (Børve, 2012). ACDC has changed name to MTE to capture the target group. ACDC is mainly based on Cognitive Behavior Theory (CBT). The techniques that individuals are taught in CBT are acknowledged as one of the most efficient interventions for preventing and reducing depression (Clarke et al., 1995; Cuijpers et al., 2009). CBT delivered as group-therapy is effective in reducing major depression (Rohde et al., 2004; Rosselló, Bernal, & Rivera-Medina, 2012). The intention is to modify dysfunctional thinking and behaviour, since these aspects are regarded as one of the main causes of depression. A depressed individual is characterised as a person who has a negative internal dialog that maintains negative experiences and beliefs (Weersing, Rozenman, & Gonzalez, 2009).

METHOD. Sample All first-year students in nine public high schools in the region of "Østfold fylkeskommune", and one school in "Akershus fylkeskommune" are implementing MTE in their ordinary school schedule. The principals for each school have choosen which classes that will attend in the study. The students in these classes are invited to attend the research project and respond to questionnaires. It is voluntary to respond. The target group is 16 and 17 years old students, irrespective of school achievements and internalizing problems. The sample consists of approximately 110 high school classes (2200 students). The classes will be randomly divided into two groups (see "Design").

Intervention. The program teaches students how to reflect about situations and their thinking-style, identify their own reaction-patterns to stressful events, to predict and influence their reactions, and to integrate this understanding and these skills into practice. Examples of themes are: how emotions emerge, how thoughts and actions influence feelings, how to change perspectives, coping techniques and how to do exercises in these methods. It combines interventions from Ellis and Grieger's (1977) Rational Emotive Behaviour Therapy (REBT) and Beck, Rush, Shaw, and Emery's (1979) cognitive behaviour therapy (CBT). In addition, MTE has elements from meta-cognition (Wells et al., 2009), positive psychology (Seligman, 2006), social theories (Bandura, 1977), mindfulness and philosophy, and modern neurobiological perspectives.

In the current project, only teachers will be course leaders and teach the students. In CWD and ACDC, course leaders have at least three years of relevant higher education; often nurses, or school-nurses, and psychologist. To be certified, the course leader in MTE, CWD and ACDC must complete a five-day intensive training program (36 hours). The organization "Fagakademiet" educates course leaders, and the training is held by a psychologist specialized in CBT. There are standardized course leader manuals and textbooks. In this project, approximately 170 teachers will be trained in MTE. The MTE course is once every week for 90 minutes across eight weeks, and have two booster sessions. After this project, the teachers will be continuing this work, because the school managements have decided to include MTE in the ordinary school plan. MTE is not treatment of mental illness.

Research questions.

The researchers hypotheses that participating in Mind power will increase self-efficacy (coping), self-esteem, self-control, quality of life and perceptions of their mental health, and reduce symptoms of anxiety and depression. The researchers want to test the effects of Mind power on school grades and drop-out. Separate analyses will be conducted on the whole intervention group vs. the control group and on the high-risk group versus the low risk group (HRG, LRG). The effects on all outcome measures will be examined after 1 year, and there will be conducted a cost-effectiveness-analysis. If more founding, the data collection will end in 2037 (the researchers have permission from The Norwegian National Research Ethics Committees). The four main hypotheses:

1. Mind power enhances school grades, self-efficacy, self-control, self-esteem, mental well-being and mental health perceptions compared to the control group.
2. Mind power prevents and reduces school dropout, and symptoms of depression and anxiety compared to the control group.
3. More cases of prevented and reduced school dropout, and symptoms of depression and anxiety are found in the LRG group than in the HRL group.
4. Gain from prevented dropouts and mental distress among LGR and HRG exceed the costs of Mind power.

Design. The design is a longitudinal randomized controlled cluster trial, where entire classes will be randomly divided into two groups. The total sample will be measured when the first group starts Mind power. The first group starts Mind power immediately, and the second group starts Mind power after six months (in the next semester). The second group functions as a control group until beginning Mind power. This delayed intervention design will allow us to differentiate between a natural increase in the outcome variables and an increase caused by Mind power, in addition to comparing two Mind power interventions at follow up. The students respond on questionnaires before the session starts on the first course day, and at the end of the sessions on the last course day (day 8), when the other group attend the course, and follow-ups. The students click on a link on iPads or Laptops when responding on the questionnaires. The design makes us able to compare the two groups, and analyze the immediate effects of MTE and the long-term effect over at least 1 year (hopefully, there will be follow-ups until 15 years, if the project receive more founding), and to test Rose's proposition that a universal strategy is more effective than a high-risk strategy.

ELIGIBILITY:
Inclusion Criteria:

* 10 high Schools have implemented Mind Power in their ordinary scheduals. We include all the students in these school classes, all the classes that the school principals have desided can attend in the study. The Principals choose which classes that will attend in the study, due to the amount of teachers who are able to attend in the project, and due the fixed time scheduals in their ordinary school plan. Then we randomize which of these school classes that starts Mind Power first (Group 1) and which starts six months later (Group 2).

Exclusion Criteria:

* none

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1673 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Hopkins Symptom Checklist (HSCL-Short form, 8 items) | 2 minutes
  Standardized and validated questionnaire: symptoms of anxiety and depression

SECONDARY OUTCOMES:
Rosenberg Self-Esteem Scale (RSES, short form, 4 items) | 1 minute
  Standaardized and validated: Self-Esteem
Lindsley self-regulation (13 items) | 2 minutes
  Standardized and validated: Self-Regulation
The Warwick-Edinburgh Mental Well-being Scale (WEMWBS, 14 items) | 2 minutes
  Standardized and validated: Mental well-being scale
The Norwegian Version of the General Perceived Self-Efficacy Scale (short form, 5 items) | 1 minute
  Standardized and validated: Self-Efficacy
Reynolds Adolescent Depression Scale, 2nd Ed. Short Form (10 items) | 1 minute
  Standardized and validated: Depression

OTHER OUTCOMES:
Students feedback on the experience of attending Mind Power | 2 minutes
  Evaluation form: with questions regarding the young people's experience of the programme in their local context.
The seven mental health rights | 4 minutes
  24 questions rearding the students belifs about the meening of life

CONTACTS AND LOCATIONS:
Overall Officials: Gry A Sælid, phd, Principal Investigator — Norwegian Institute of Public Health
Locations (1):
- Gry Anette Sælid, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Services of sensitiv data (TSD) at the University of Oslo is providing this option.

REFERENCES:
- [Derived] Saelid GA, Czajkowski NO, Aaro LE, Andersen JR, Idsoe T, Helleseter MD, Holte A. Effects of a school-based intervention on levels of anxiety and depression: a cluster-randomized controlled trial of the MindPower program in ten high schools in Norway. BMC Psychol. 2022 Jan 24;10(1):14. doi: 10.1186/s40359-022-00721-y. PMID 35074007